CLINICAL TRIAL: NCT05264922
Title: Stromal Vascular Fraction (SVF) Cells for Non-Operative Treatment of Small Rotator Cuff Tears
Acronym: SVF
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never started. PI left institution.
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1719310
Record Dates: First submitted 2021-12-27; First posted 2022-03-03 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to SVF Cells & Fibrin Glue or Fibrin Glue alone.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The provider (PI) and team performing the injection will not care for the subject during follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fibrin Glue (Active Comparator): Single 4 milliliter (mL) injection of 0.9% normal saline and fibrin glue solution
  Interventions: Drug: Tisseel Injectable Product
- SVF cells and Fibrin Glue (Experimental): Nucleated adipose-derived cells loaded in a fibrin glue scaffold
  Interventions: Drug: Tisseel Injectable Product; Biological: Stromal Vascular Fraction Cells

INTERVENTIONS:
Drug: Tisseel Injectable Product — Fibrin glue will provide an inert, biocompatible, viscous substance able to remain within the Rotator Cuff (RC) defect rather than injecting SVF cells in saline.
  Other Names: Fibrin Glue
Biological: Stromal Vascular Fraction Cells — Stromal Vascular Fraction cells are autologously harvested, processed and reinjected into the affected shoulder.
  Arms: SVF cells and Fibrin Glue

SUMMARY:
The investigator's goal is to determine the effectiveness of stromal vascular fraction (SVF) cell injection to treat small rotator cuff tears without surgery.

DETAILED DESCRIPTION:
Small rotator cuff tendon tears are a hard task in shoulder care. They are often not operated on because research has not shown any increased benefit of surgery over physical therapy. The most common way to treat these tears is through physical therapy or steroid injections. However, the relief doesn't last very long. Recent studies have shown a lot of tears get worse over time. This happens because the physical therapy options can treat the pain and symptoms, but do not heal the actual tear.

Another non-surgical option for treating small tears is through adipose-derived stem cells. Adipose-derived stem cells are cells that are found in the fat in our bodies. The cells have shown promise in fixing tissues and may provide help to treat small rotator cuff tears. The investigators are studying a part of these fat cells known as the stromal vascular fraction (SVF). The SVF contains a number of cells that are able to become a variety of different cells. This is important because they may be able to turn into cells that may help heal the damaged rotator cuff tendons. These cells have been shown to improve results after rotator cuff surgery, but no research has used these cells to help small tears without surgery. The use of SVF is investigational. "Investigational" means that the drug being tested has not been approved for routine clinical use or for the use described in this study by the United States Food and Drug Administration (FDA). The FDA is allowing the use of this drug for research. The investigators goal is to determine the effectiveness of SVF cell injection to treat small rotator cuff tears without surgery.

ELIGIBILITY:
Inclusion Criteria

1. Male and female patients 30-65 years of age
2. Symptomatic partial-thickness rotator cuff tears
3. Suitable candidate for lipoaspiration and autologous adipose derived stem cell therapy as per physician.

Exclusion Criteria

1. History of RC repair of affected shoulder, osteomyelitis or septic arthritis;
2. Primary diagnosis of osteoarthritis, primary adhesive capsulitis;
3. Full thickness rotator cuff tear
4. RC tear of the subscapularis (SSc) or teres minor (TM), or a RC tear at the musculotendinous junction.
5. Prescribed physical therapy or injection (of any nature) to shoulder prior to initial visit (within past 3 months);
6. Clinically significant medical diseases that can impact tissue healing (i.e. Cardiovascular/peripheral vascular disease, diabetes, cancer, endocrine disease, hepatic disease (hepatitis), renal disease, autoimmune/inflammatory disease, HIV;
7. Cervical spine radiculopathy;
8. Current anticoagulation therapy (excluding Aspirin 81mg), immunosuppressant medication, narcotic use;
9. Women of child bearing potential must test negative on standard urine pregnancy test and must agree to practice appropriate contraception for the first year of the study (i.e. oral contraceptive, barrier method, intrauterine device (IUD), intramuscular contraceptive);
10. Subjects with abnormal hematology or serum chemistry lab results, outside of the normal range, as defined by the American Board of Internal Medicine (ABIM) Laboratory Test Reference Ranges, which are clinically significant, in the opinion of the investigator;
11. BMI greater than 40 kg/m2;
12. History of tobacco use within last 3 years;
13. Subject has been diagnosed with any bleeding disorders, including but not limited to: hemophilia A or B, Von Willebrand Disease;
14. Currently participating, or has participated in any other clinical trials within 6 months prior to the screening visit;
15. Subjects has any significant medical condition, that in the option of the investigator, would make them unable to provide informed consent and/or interfere with their compliance of study requirements;
16. Subject has a documented allergy to the anesthetic or any component of the injectable, including but not limited to: aprotinin.
17. Subject has a contraindication for completing the MRI (i.e. pacemaker, aneurysm clip, metal fragments, etc that may become dislodged) or has problems with loud noises or claustrophobia.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-09 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy - MRI-measured healing rate in the rotator cuff tear | 24 months
  Healing rates between the treatment with stromal vascular fraction (SVF) cells and exercise program (EP) group will be compared to the sham and EP group.
Primary Safety - Incidence/Rates of adverse events (AEs) involving the affected joint | 24 months
  Both study-related AE assessments and the clinical record will be interrogated to determine if the subjects had any adverse events involving the affected joint. Incidence and rates of AEs between the treatment with stromal vascular fraction (SVF) cells and exercise program (EP) group will be compared to the sham and EP group.

SECONDARY OUTCOMES:
Patient-reported measures Western Ontario Rotator Cuff (WORC) Index | 24 months
  WORC score - Compare clinical outcomes between treatment with stromal vascular fraction (SVF) cells and EP and sham injection and EP. The investigators expect the SVF-treated patients to improve by over 12% on the WORC at the final 2-yr follow-up.
Patient-reported measures Patient Reported Outcomes Measurement Information System (PROMIS) | 24 months
  PROMIS score - Compare clinical outcomes between treatment with stromal vascular fraction (SVF) cells and EP and sham injection and EP.expect the SVF-treated patients to improve by 10 points on the PROMIS at the final 2-yr follow-up.
Patient-reported measures Visual Analog Scale (VAS) | 24 months
  Pain VAS score - Compare clinical outcomes between treatment with stromal vascular fraction (SVF) cells and EP and sham injection and EP. expect the SVF-treated patients to improve by over 12% on the WORC, by 10 points on the PROMIS, and by 20% on the pain VAS by the final 2-yr follow-up. expect the SVF-treated patients to improve by 20% on the pain VAS at the final 2-yr follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Awan, DO, Principal Investigator — AdventHealth Orlando
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No